CLINICAL TRIAL: NCT05040490
Title: Comparison of the Effects of Neostigmine and Sugammadex on Postoperative Residual Curarization and Postoperative Pulmonary Complications Detected by Diaphragm and Lung Ultrasonography: A Study Protocol for Prospective Double-blind Randomized Controlled Trial.
Brief Title: Influence of Neostigmine vs. Sugammadex on PORC and PPCs by Ultrasonography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jie YI, deputy director of surgery department, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Diaphragm/Lung Ultrasound
Record Dates: First submitted 2021-08-25; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pulmonary Complications
Keywords: postoperative pulmonary complications; postoperative residual curarisation; lung ultrasound; diaphragm ultrasonography
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUG group (Experimental): sugammadex as reversal drugs
  Interventions: Drug: sugammadex as reversal drugs
- NEO group (No Intervention): neostigmine as reversal drugs

INTERVENTIONS:
Drug: sugammadex as reversal drugs — use sugammadex to reverse neuromuscular blockade
  Arms: SUG group

SUMMARY:
This trial aims to compare the incidence of postoperative residual curarisation (PORC) and postoperative pulmonary complications (PPCs) in the SUG and NEO group by means of diaphragm ultrasonography and LUS, so as to conclude whether SUG can outperform NEO in preventing occurrence of PORC and PPCs.

DETAILED DESCRIPTION:
The incidence of postoperative residual curarisation (PORC) is about 2%-64% worldwide, which may be an underling risk factor of postoperative pulmonary complications (PPCs), causing many undesirable effects on patients. Thus, reversal drugs of neuromuscular blocking agents (NMBAs) such as neostigmine (NEO) and sugammadex (SUG) have been administrated, and SUG maybe perform better in preventing PORC. Different supplementary methods to help identify PORC or PPCs have also been reported, such as adductor of pollicis acceleromyography and lung ultrasound (LUS). Recently, diaphragm ultrasonography has been used to evaluate PORC, as a novel approach.In this prospective, double-blind, randomized controlled trial, we will enroll 414 patients of American Society of Anesthesiologists physical status I-III, aged over 60 years, who will be scheduled to undergo arthroplasty surgery under general anesthesia. Participants will be randomized into NEO and SUG group receiving neostigmine and sugammadex as reversal drug respectively. The primary outcomes will be the incidence of PPCs in NEO and SUG group respectively. The secondary outcome is the incidence of PORC in the two groups.We hypothesize that: 1) the incidence of PPCs is lower after reversal with SUG than with NEO, 2) using the method of diaphragm ultrasonography, the incidence PORC is lower after reversal with SUG than with NEO, 3) the incidence of PPCs can be predicted by LUS and by evaluating whether there is PORC through diaphragmatic ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status I-III
2. Aged over 60 years
3. Anesthesia induction with rocuronium as NMBAs, maintenance with volatile sevoflurane
4. Scheduled to undertake joint surgery
5. Signed the informed consent form

Exclusion Criteria:

1. Those with a history of hepatic or renal disease, chronic or acute alcoholism, allergy or hypersensitivity to sugammadex or neostigmine, current medication with effects on the central nervous system, a history of dysfunction of neuromuscular system
2. Those with diaphragm insufficiency or massive pleural effusion
3. Women who are pregnant or nursing
4. Those undergoing upper abdominal laparotomy, after which we cannot obtain a satisfactory ultrasound imaging or do not have space for placement of ultrasonic probe
5. Declined to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2021-08-31 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative pulmonary complications | 30 days after surgery
  incidence of postoperative pulmonary complications

SECONDARY OUTCOMES:
Evaluation of diaphragmatic and pulmonary function by means of diaphragm and lung ultrasonography | preoperatively, 10min and 30min after extubation for diaphragm ultrasonography and LUS
  Evaluation of diaphragmatic and pulmonary function by means of diaphragm and lung ultrasonography(LUS)

OTHER OUTCOMES:
sedation score | 10min and 30min after extubation
  sedation score OAAS
duration of hospitalization | 30 days after surgery
  duration of hospitalization
dosage of intravenous and inhaling sedative drug, analgesia drug, NMBAs | 30 days after surgery
  dosage of intravenous and inhaling sedative drug, analgesia drug, NMBAs
duration of surgery and anesthesia | 30 days after surgery
  duration of surgery and anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: ZHANG YUGUAN, doctoral, Principal Investigator — Peking Union Medical College Hospital

REFERENCES:
- [Derived] Zhang YG, Chen Y, Zhang YL, Yi J. Comparison of the effects of neostigmine and sugammadex on postoperative residual curarization and postoperative pulmonary complications by means of diaphragm and lung ultrasonography: a study protocol for prospective double-blind randomized controlled trial. Trials. 2022 May 7;23(1):376. doi: 10.1186/s13063-022-06328-3. PMID 35526047